CLINICAL TRIAL: NCT03297099
Title: A Prospective Cohort Study: Robotic-Assisted Laparoscopic Versus Open Surgery for Complicated Hepatolithiasis
Brief Title: Robotic-Assisted Laparoscopic Versus Open Surgery for Complicated Hepatolithiasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Shuguo Zheng, MD, Professor of Hepatobiliary Surgery Institute; Chief Physician; Administrator of laparoscopic department, Southwest Hospital, China
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SWHZSG006; Zhengshuguo (Registry Identifier: Zhengshuguo)
Record Dates: First submitted 2017-09-21; First posted 2017-09-29 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Hepatolithiasis
Keywords: robot-assisted laparosocpic; hepatectomy
MeSH Terms: interventions — Conversion to Open Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robot-assisted Laparoscopic operation (Experimental): Da Vinci surgical robot can overcome limitations of conventional laparoscopic surgery in terms of vision and instrumentation flexibility, making the minimally invasive treatment of complex hepatolithiasis possible.
  Interventions: Procedure: Robot-assisted Laparoscopic operation
- Open surgery (Active Comparator): The indication of laparoscopic surgery is mainly for early regional type hepatolithiasis. Open surgery is the traditional treatment method for heptolithiasis.
  Interventions: Procedure: open surgery

INTERVENTIONS:
Procedure: Robot-assisted Laparoscopic operation — Thirty patients with hepatolithiasis were selected and divided into robot group as described in the detailed description. Under general anesthesia, the patient was placed in a supine 30-degree reverse Trendelengburg position with both legs separating. The surgeon work on the console, and assist surgeon stand between legs. Operation began with division of liver ligaments, liver mobilization, followed by intrahepatic access to the Glissonian pedicle . A endoscopic stapler devices was used for Glissonian pedicle cutting and suture. Liver parenchyma was divided by harmonic scalpel combined with vascular stapler.
  Arms: Robot-assisted Laparoscopic operation
Procedure: open surgery — surgery group as described in the detailed description.Open surgery was performed under general anesthesia with the patient in the supine position. Routinely, a reversed L-shape incision was performed. Operation began with division of liver ligaments, liver mobilization, followed by intrahepatic access to the Glissonian pedicle . A endoscopic stapler devices was used for Glissonian pedicle cutting and suture. Liver parenchyma was divided by harmonic scalpel combined with vascular stapler.
  Arms: Open surgery

SUMMARY:
The indication of laparoscopic surgery is mainly for early regional type hepatolithiasis. Open surgery is the traditional treatment method for heptolithiasis. Da Vinci surgical robot can overcome limitations of conventional laparoscopic surgery in terms of vision and instrumentation flexibility, making the minimally invasive treatment of complex hepatolithiasis possible. The study aimed to evaluate the safety, feasibility, and efficacy of robot assist laparoscopic surgery for the treatment of complicated hepatolithiasis by contrast of open procedures.

DETAILED DESCRIPTION:
Robot-assisted laparoscopic operation is a safe and feasible treatment for selected patients with complicated hepatolithiasis, with an advantage over open surgery in the field of intraoperative blood loss, less hilar occlusion, lower transfusion rate, less postoperative hospital stay.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with intrahepatic bile duct stones or hepatolithiasis.
2. Liver function > Child-pugh level B, no severe biliary cirrhosis, ICG ≤ 15%, the residual liver volume and standard liver volume ratio ≥ 40%. The conditions of open hepatectomy were achieved
3. Age: Between 18 to 70 years
4. Combined with severe liver atrophy hypertrophy syndrome, hepatic portal transposition or hilar biliary fibrosis / stenosis
5. Patients with good general condition, the conditions of open Anatomical Hepatectomy were achieved
6. Other organ lesions and previous biliary tract operation is not the absolute exclusion criteria
7. Written informed consent

Exclusion Criteria:

1. Patients with bad general condition or important organ lesions, liver resection could not be tolerated
2. Age:Younger than 18 or more than 70 years old
3. Malignant tumor recurrence within one month postoperation
4. Complicated case need to get emergency operation
5. Contraindication of laparoscopy: Combined with complicated acute cholangitis, repeated biliary tract operation, heavy intra-abdominal adhesion, Trocar can not be placed in. Artificial pneumoperitoneum could not be tolerated

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
initial stone clearance rate | during the operation
  rate of the removal of the stones from intrahepatic bile duct identified by ultrasonic or computed tomography or magnetic resonance

SECONDARY OUTCOMES:
intraoperative parameters | during the operation
  operation time, intraoperative blood loss, rate of blood transfusion

OTHER OUTCOMES:
postoperative complications | Duration hospitalization(an expected average of 7 days)
  ascites, pleural effusion,cardiopulmonary insufficiency,mortality, postoperative liver function failure.

CONTACTS AND LOCATIONS:
Overall Officials: Shuguo Zheng, Study Director — Shuguo Zheng, MD Study Director Institute of Hepatobiliary Surgery ,Southwest Hospital ,Third Military Medical University
Locations (1):
- Southwest Hospital, Chongqing, Chongqing Municipality, China